CLINICAL TRIAL: NCT00915876
Title: Effects of 19-nor-1α-dihydroxyvitamin D2 (Paricalcitol) Versus Placebo on Oxidative Stress and Vascular Reactivity in CKD Patients
Brief Title: Vascular Reactivity in Chronic Kidney Disease (CKD) Patients Receiving Paricalcitol Versus Placebo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amy Barton Pai (Other)
Collaborators: Albany College of Pharmacy and Health Sciences (Other)
Responsible Party: Sponsor-Investigator, Amy Barton Pai, Associate Professor, University of Michigan
Organization: University of Michigan (Other)
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: Paricalcitol-AMC2443
Record Dates: First submitted 2009-06-05; First posted 2009-06-08 (Estimated); Results first posted 2016-12-02 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Kidney Disease
Keywords: chronic kidney disease; Vitamin D
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — paricalcitol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paricalcitol (Active Comparator)
  Interventions: Drug: Paricalcitol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Paricalcitol — paricalcitol 1 mcg QD x 8 weeks
  Arms: Paricalcitol
Drug: Placebo — Placebo for Paricalcitol 1 mcg QD x 8 weeks
  Arms: Placebo

SUMMARY:
This research is studying how Vitamin D may affect blood vessels reaction to stress and blood levels of substances that may increase blockages in the blood vessels in chronic kidney disease (CKD) patients. Blood vessel health is worsened in CKD and some studies have shown that Vitamin D improves blood vessel health. The type of Vitamin D being used in this study (paricalcitol) is Food and Drug Administration (FDA) approved to treat high parathyroid hormone levels. The purpose of this study is to find out if paricalcitol has other benefits beyond its ability to lower parathyroid hormone levels such as improving the blood vessels reaction to stress and decreasing blood levels of substances that may increase blockages in the blood vessels.

ELIGIBILITY:
Inclusion Criteria:

* Males or females ≥ 18 years of age at the start of screening
* CKD with eGFR 15-60 mL/min/1.73m2 by MDRD
* Not expected to start dialysis for 4 months
* Serum intact PTH 70-200 pg/mL during screening period
* On stable ACEI/ARB regimen for 30 days prior to screening

Exclusion Criteria:

* History of any of the following diseases:

  * congestive heart failure
  * MI within the last 6 months
  * history of cerebrovascular accident
  * significant valvular disease
  * malignancy
* Currently taking any vitamin D products
* Mean systolic blood pressure values > 190 or diastolic blood pressure values > 100 mm/Hg during the preceding 30 day period prior to screening
* Currently being titrated on therapy with an angiotensin converting enzyme inhibitor or angiotensin receptor blocker
* Two consecutive serum calcium values greater than 10.2 mg/dL or Ca x P > 55 mg2/dL2
* Currently receiving erythropoiesis stimulating agent or intravenous iron therapy
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Pai, Pharm.D., Principal Investigator — Albany College of Pharmacy and Health Sciences; Amy Pai, PharmD, Principal Investigator — Albany College of Pharmacy and Health Sciences
Locations (1):
- Albany Medical Center South Clinical Campus, Albany, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Paricalcitol | Placebo
Started | 20 | 21
Moving Beyond First Dose | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: One placebo group patient dropped out due to an adverse event is not included in baseline measures or in outcome measures. Assuming 35% variability in circulating ICAM-1 concentrations,46 a sample size of 18 per group is adequate to detect a 50 percentage point difference in the percent in ICAM-1 with 80% power and an = 0.05.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Paricalcitol | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (11) | 64 (14) | 66 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 12 | 19
  Male | 13 | 8 | 21
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40
estimated glomerular filtration rate [Mean (Standard Deviation); unit: mL/min/1.73m2] | 36 (11) | 30 (9) | 35 (10)

OUTCOME MEASURES:

1. Primary Outcome: Change in Circulating ICAM-1 Shown by Absolute Values at Baseline, Day 28 and Day 56
Description: Values of ICAM-1 (intracellular adhesion molecule) a measure of vascular reactivity, at three time points: baseline, day 28, and day 56
Time Frame: Day 28 and Day 56
Measure: Mean (Standard Deviation); unit: nanogram/ml
Arm/Group | Placebo | Paricalcitol
Number analyzed (Participants) | 20 | 20
nanogram/ml
  Baseline | 707 (504) | 701 (603)
  Day 28 | 679 (557) | 627 (570)
  Day 56 | 590 (458) | 477 (382)
Statistical Analysis 1: Comparison: Placebo vs Paricalcitol; Test type: Superiority or Other; p > 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: TENTATIVE: 7 weeks of intervention and 30 days of followup, totalling up to 12 weeks per person
Arm/Group | Placebo | Paricalcitol
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 1/21 | 0/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=21) | Paricalcitol (N=20)
Weakness (Nervous system disorders) | 1 (1) | 0 (0) — Patient took one dose of placebo and complained of weakness. The study drug was stopped and the dose of gabapentin the patient was taking was higher than recommended for his renal function which was addressed by the attending physician.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No